CLINICAL TRIAL: NCT01686477
Title: Preterm Formula or Donor Breast Milk to Make up Any Shortfall in Mother's Own Milk
Brief Title: PREterM FOrmula Or Donor Breast Milk for Premature Babies
Acronym: PREMFOOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRO2006
Record Dates: First submitted 2012-08-07; First posted 2012-09-18 (Estimated); Results first posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2023-10

CONDITIONS: Adiposity; Insulin Resistance; Metabolomic Profile; microRNA Profile
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Unfortified Human Donor Milk (Active Comparator): Used to make up any shortfall in mother's own milk
  Interventions: Other: Unfortified Human donor Milk used to make up any shortfall in mother's own milk
- Fortified Human Donor Milk (Active Comparator): Used to make up any shortfall in mother's own milk
  Interventions: Other: Fortified Human donor Milk used to make up any shortfall in mother's own milk
- Preterm Formula (Active Comparator): Used to make up any shortfall in mother's own milk
  Interventions: Other: Preterm Formula used when there is a shortfall in mother's own milk

INTERVENTIONS:
Other: Unfortified Human donor Milk used to make up any shortfall in mother's own milk
  Arms: Unfortified Human Donor Milk
Other: Fortified Human donor Milk used to make up any shortfall in mother's own milk
  Arms: Fortified Human Donor Milk
Other: Preterm Formula used when there is a shortfall in mother's own milk
  Arms: Preterm Formula

SUMMARY:
In order to address this crucial question, central to preterm newborn care, a multicentre United Kingdom (UK) -wide study randomising 4000 preterm babies would be necessary to achieve sufficient power to evaluate the impact on the short-term outcomes necrotising enterocolitis and bloodstream infection, and establish cohorts large enough to address long-term metabolic (such as obesity, type 2 diabetes), cardiovascular (such as blood pressure) and developmental outcomes. This pilot trial will evaluate the practicability and feasibility of such a large multicentre UK randomised controlled trial. In addition to evaluating feasibility and to ensure maximal use of resources allocated, this study will also assess outcomes that are indicative of long term metabolic health.

DETAILED DESCRIPTION:
Mother's Own Milk (MOM) is recommended for preterm babies. However, on average, mothers giving birth preterm are able to provide less than half their baby's milk requirements. Standard clinical practice is to make up any shortfall in MOM with either pasteurised Human Donor Milk (HDM) or Preterm Formula (PTF). Which option is more beneficial to clinical outcomes is unknown.

Pasteurisation reduces or destroys many biologically active components and HDM, unlike PTF, is very variable in composition. Clinicians who use HDM do so primarily in the hope that despite pasteurisation it will reduce bloodstream infection and necrotising enterocolitis, a serious, devastating inflammatory disease characterised by bowel death and multisystem failure. These are two of the most feared conditions in newborn medicine as described above. Landmark nutritional trials in the early 1980's suggest positive effects of human milk on insulin sensitivity, and other metabolic outcomes. Clinicians who prefer PTF believe it benefits growth, including brain growth, and improves neurodevelopmental outcome.

Neonates born below 32 weeks gestational age will be randomised to receive fortified HDM, unfortified HDM, or PTF to make up any shortfall in MOM until 35 weeks postmenstrual age with a sample size of 22 in each group. The trial is designed to reflect current preterm feeding practice. The trial will take place in neonatal units in London and parent consent obtained within 48hr of birth. Permission will be sought for long term follow up, initially from parents (later from children themselves). Outcomes will be body composition using magnetic resonance imaging and other imaging techniques. This pilot study will specifically assess feasibility by testing 1) provision of HDM by Human Milk Banks in London 2) acceptability to parents and clinicians using feedback on trial design 3) recruitment to target and 4) retrieval of clinical data for all recruited babies form the National Neonatal Database.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born between 25+0 to 31+6 weeks gestational age
* Written informed consent from parents

Exclusion Criteria:

* Major congenital or life threatening abnormalities or congenital abnormalities that preclude early milk feeding
* Inability to randomise infant within 48 hours

Ages: 25 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2013-04-02 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neena Modi, MBChB, Principal Investigator — Imperial College London
Locations (1):
- Chelsea and Westminster Hospital Neonatal Unit, London, United Kingdom

REFERENCES:
- [Derived] Quigley M, Embleton ND, Meader N, McGuire W. Donor human milk for preventing necrotising enterocolitis in very preterm or very low-birthweight infants. Cochrane Database Syst Rev. 2024 Sep 6;9(9):CD002971. doi: 10.1002/14651858.CD002971.pub6. PMID 39239939

RESULTS

PARTICIPANT FLOW:
Groups:
- Unfortified Human Donor Milk: Used to make up any shortfall in mother's own milk
  Unfortified Human donor Milk used to make up any shortfall in unfortified mother's own milk
- Fortified Human Donor Milk: Used to make up any shortfall in mother's own milk
  Fortified Human donor Milk used to make up any shortfall in fortified mother's own milk
- Preterm Formula: Used to make up any shortfall in mother's own milk
  Preterm Formula used when there is a shortfall in mother's own milk
Period: Feeding Intervention
Arm/Group | Unfortified Human Donor Milk | Fortified Human Donor Milk | Preterm Formula
Started | 35 | 34 | 34
Completed | 32 | 25 | 31
Not Completed | 3 | 9 | 3
Not completed — Death | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 6 | 0
Not completed — Physician Decision | 1 | 2 | 0
Not completed — Met pre-defined safety threshold | 1 | 0 | 1
Not completed — Transfer to a non-participating hospital | 0 | 1 | 1
Period: Primary Outcome Term Scan
Arm/Group | Unfortified Human Donor Milk | Fortified Human Donor Milk | Preterm Formula
Started | 30 (32 completed feed intervention; 28 completed feed intervention and consented to scans; 2 not completed feed intervention but consented to scans) | 25 (25 completed feed intervention; 22 completed feed intervention and consented to scans; 3 not completed feed intervention but consented to scans) | 30 (31 completed feed intervention; 28 completed feed intervention and consented to scans; 2 not completed feed intervention but consented to scans)
Completed | 21 | 19 | 24
Not Completed | 9 | 6 | 6
Not completed — Withdrawal by Subject | 6 | 5 | 5
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Scanner unavailable to measure primary outcome | 2 | 0 | 0
Period: Term Plus 6 Week Scan (End of Study)
Arm/Group | Unfortified Human Donor Milk | Fortified Human Donor Milk | Preterm Formula
Started | 21 | 19 | 24
Completed | 14 (13 completed feed intervention and consented to scans; 1 not completed feed intervention but consented to scans) | 5 (5 completed feed intervention and consented to scans) | 19 (18 completed feed intervention and consented to scans; 1 not completed feed intervention but consented to scans)
Not Completed | 7 | 14 | 5
Not completed — Withdrawal by Subject | 7 | 12 | 5
Not completed — Lost to Follow-up | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Unfortified Human Donor Milk: Used to make up any shortfall in mother's own milk
  Unfortified Human donor Milk used to make up any shortfall in mother's own milk
- Fortified Human Donor Milk: Used to make up any shortfall in mother's own milk
  Fortified Human donor Milk used to make up any shortfall in mother's own milk
- Total: Total of all reporting groups
Arm/Group | Unfortified Human Donor Milk | Fortified Human Donor Milk | Preterm Formula | Total
Number analyzed (Participants) | 35 | 34 | 34 | 103
Age, Continuous [Mean (Standard Deviation); unit: Completed gestational weeks] — Completed gestational weeks (decimal)
  Completed gestational weeks | 29.4 (2.2) | 29.6 (2.0) | 29.7 (1.7) | 29.5 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 15 | 43
  Male | 20 | 21 | 19 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 35 | 34 | 34 | 103
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 35 | 34 | 34 | 103

OUTCOME MEASURES:

1. Primary Outcome: Total Body Adiposity
Description: As measured by whole body Magnetic Resonance Imaging (MRI). MR images were acquired using a rapid T1-weighted spin-echo sequence allowing whole body imaging. Images obtained give good contrast between adipose tissue and other tissues, and allows direct measurement of adipose compartment volumes, whole body adipose volume being the sum of these compartments. The time taken to reach term age equivalent will vary depending on the birth gestational age of the infant. The range will be 8-15 weeks (representing gestational birth age from 25-32 weeks).
Time Frame: Measured as close as possible to the baby's due date, at an average age of 10 weeks (range 8 to 15 weeks)
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Unfortified Human Donor Milk | Fortified Human Donor Milk | Preterm Formula
Number analyzed (Participants) | 21 | 19 | 24
Litres | 0.893 (0.38) | 0.863 (0.26) | 0.809 (0.25)

2. Secondary Outcome: Consent Rate for Feeding Intervention (Opt Out Approach)
Description: Consent rate for feeding intervention of number of parents of eligible infants approached and study discussed with (opt out approach)
Time Frame: Up to the first 48hrs of life
Population: Parents of 165 eligible infants for which the study was discussed with and opportunity offered to opt-out from randomisation to feed intervention
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Opt out consent for feed intervention
Arm/Group | All Participants
Number analyzed (Participants) | 165
Participants | 103

3. Secondary Outcome: Parental Withdrawal From Feed Intervention
Description: Parental withdrawal rate from feed intervention
Time Frame: From birth to 35 weeks post menstrual age
Population: All participants
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: All participants
Arm/Group | All Participants
Number analyzed (Participants) | 103
Participants | 6

4. Secondary Outcome: Parental Withdrawal Rate From Feed Intervention by Arm
Description: Parental withdrawal rate from feed intervention by feed intervention arm
Time Frame: From birth to 35 weeks post menstrual age
Population: Parental withdrawal rate from feed intervention by arm
Measure: Count of Participants; unit: Participants
Groups:
- Unfortified Human Donor Milk: Unfortified Human Donor Milk Feed Intervention Arm
- Fortified Human Donor Milk: Fortified Human Donor Milk Feed Intervention Arm
- Preterm Formula: Preterm Formula Feed Intervention Arm
Arm/Group | Unfortified Human Donor Milk | Fortified Human Donor Milk | Preterm Formula
Number analyzed (Participants) | 35 | 34 | 34
Participants | 0 | 6 | 0

5. Secondary Outcome: Clinician Refusal to Randomise
Description: Attending clinician refusal to randomise eligible infant into feeding intervention
Time Frame: Up to the first 48hrs of life.
Population: All eligible participants who consented for feed intervention who were then not randomised due to clinician refusal
Measure: Count of Participants; unit: Participants
Groups:
- All Eligible Participants Who Consented for Feed Intervention: All eligible participants who consented for feed intervention who were then not randomised due to clinician refusal
Arm/Group | All Eligible Participants Who Consented for Feed Intervention
Number analyzed (Participants) | 103
Participants | 0

6. Secondary Outcome: Safety Criteria Threshold
Description: Number of infants who met the weight gain safety criteria. Safety criteria defined by slow growth were based on the UK Neonatal and Infant Close Monitoring growth chart 2009: if after two weeks of reaching a milk volume of 120ml/kg/d, the infant showed a 3 marked centile downward crossing (equating to approximately a 1.4-2.0 z-score change from birthweight) fortification or formula was commenced
Time Frame: Birth to 35 weeks post menstrual age
Population: All participants who consented for feed intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Unfortified Human Donor Milk | Fortified Human Donor Milk | Preterm Formula
Number analyzed (Participants) | 35 | 34 | 34
Participants | 1 | 0 | 1

7. Secondary Outcome: Weight at Term
Description: Weight at term by feed intervention arm
Time Frame: Measured as close as possible to the baby's due date, at an average age of 10 weeks (range 8 to 15 weeks)
Measure: Mean (Standard Deviation); unit: Grams
Groups:
- Unfortified Human Donor Milk: Unfortified Human Donor Milk
- Fortified Human Donor Milk: Fortified Human Donor Milk
- Preterm Formula: Preterm Formula
Arm/Group | Unfortified Human Donor Milk | Fortified Human Donor Milk | Preterm Formula
Number analyzed (Participants) | 21 | 19 | 24
Grams | 3295 (798) | 3185 (678) | 3153 (656)

8. Secondary Outcome: Length at Term
Description: Length at term by feed intervention arm
Time Frame: Term corrected age (as close as possible to due date)
Population: Feed intervention arm
Measure: Mean (Standard Deviation); unit: Cm
Arm/Group | Unfortified Human Donor Milk | Fortified Human Donor Milk | Preterm Formula
Number analyzed (Participants) | 21 | 19 | 24
Cm | 50.0 (3.8) | 49.5 (3.0) | 49.6 (3.5)

9. Secondary Outcome: Head Circumference at Term
Description: Head circumference at term by feed intervention arm
Time Frame: Term corrected age (as close as possible to due date)
Population: Feed intervention arm
Measure: Mean (Standard Deviation); unit: Cm
Arm/Group | Unfortified Human Donor Milk | Fortified Human Donor Milk | Preterm Formula
Number analyzed (Participants) | 21 | 19 | 24
Cm | 35.9 (2.4) | 35.0 (1.9) | 35.4 (2.1)

10. Secondary Outcome: Regional Adiposity, as Measured by Whole Body MRI, at Term.
Description: Internal Abdominal Adipose Tissue at Term reported here. As measured by whole body Magnetic Resonance Imaging (MRI). MR images were acquired using a rapid T1-weighted spin-echo sequence allowing whole body imaging. Images obtained give good contrast between adipose tissue and other tissues, and allows direct measurement of adipose compartment volumes. These adipose compartments are defined as superficial subcutaneous, deep subcutaneous, and internal. Each of these three compartments are further subdivided into abdominal and non-abdominal.
Time Frame: Measured as close as possible to the baby's due date, at an average age of 10 weeks (range 8 to 15 weeks)
Population: Feed intervention arm
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Unfortified Human Donor Milk | Fortified Human Donor Milk | Preterm Formula
Number analyzed (Participants) | 21 | 19 | 24
Litres | 0.043 (0.02) | 0.044 (0.02) | 0.040 (0.01)

11. Secondary Outcome: Non Adipose Tissue, as Measured by Whole Body MRI, at Term
Description: Non adipose tissue, as measured by whole body Magnetic Resonance Imaging (MRI) at term. MR images were acquired using a rapid T1-weighted spin-echo sequence allowing whole body imaging. Images obtained give good contrast between adipose tissue and other tissues, and allows direct measurement of adipose compartment volumes, whole body adipose tissue volume being the sum of these adipose compartment volumes. This volume may be converted to adipose tissue mass on the assumption that the density of adipose tissue is 0.9 g/cm³. Non adipose tissue mass reported here is weight (g) minus whole body adipose mass (g)
Time Frame: Measured as close as possible to the baby's due date, at an average age of 10 weeks (range 8 to 15 weeks)
Population: Feed intervention arm
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Unfortified Human Donor Milk | Fortified Human Donor Milk | Preterm Formula
Number analyzed (Participants) | 21 | 19 | 24
Grams | 2511.79 (502.84) | 2385.74 (437.81) | 2424.70 (462.63)

12. Secondary Outcome: Weight at Term Plus 6 Weeks
Description: Weight at Term plus 6 weeks by feed intervention arm
Time Frame: Term plus 6 weeks corrected age
Population: Feed intervention arm
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Unfortified Human Donor Milk | Fortified Human Donor Milk | Preterm Formula
Number analyzed (Participants) | 14 | 5 | 19
Grams | 4564 (982) | 4594 (802) | 4590 (820)

13. Secondary Outcome: Length at Term Plus 6 Weeks
Description: Length at Term plus 6 weeks by feed intervention group
Time Frame: Term plus 6 weeks
Population: Feed intervention arm
Measure: Mean (Standard Deviation); unit: Cm
Arm/Group | Unfortified Human Donor Milk | Fortified Human Donor Milk | Preterm Formula
Number analyzed (Participants) | 14 | 5 | 19
Cm | 55.70 (3.46) | 55.86 (2.87) | 55.98 (3.70)

14. Secondary Outcome: Head Circumference at Term Plus 6 Weeks
Description: Head circumference at Term plus 6 weeks by feed intervention arm
Time Frame: Term plus 6 weeks
Population: Feed intervention arm
Measure: Mean (Standard Deviation); unit: Cm
Arm/Group | Unfortified Human Donor Milk | Fortified Human Donor Milk | Preterm Formula
Number analyzed (Participants) | 14 | 5 | 19
Cm | 38.76 (2.13) | 37.89 (1.97) | 38.91 (2.00)

15. Secondary Outcome: Total Body Adiposity at Term Plus 6 Weeks
Description: As measured by whole body Magnetic Resonance Imaging (MRI). MR images were acquired using a rapid T1-weighted spin-echo sequence allowing whole body imaging. Images obtained give good contrast between adipose tissue and other tissues, and allows direct measurement of adipose compartment volumes, total body adipose tissue volume being the sum of all these compartment volumes.
Time Frame: Term plus 6 weeks
Population: Feed Intervention Arm
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Unfortified Human Donor Milk | Fortified Human Donor Milk | Preterm Formula
Number analyzed (Participants) | 14 | 5 | 19
Litres | 1.355 (0.486) | 1.474 (0.463) | 1.353 (0.284)

16. Secondary Outcome: Regional Adiposity, as Measured by Whole Body MRI at Term Plus 6 Weeks
Description: Regional adiposity, as measured by whole body MRI at Term plus 6 weeks, Internal Abdominal Adipose Tissue reported here. As measured by whole body Magnetic Resonance Imaging (MRI). MR images were acquired using a rapid T1-weighted spin-echo sequence allowing whole body imaging. Images obtained give good contrast between adipose tissue and other tissues, and allows direct measurement of adipose compartment volumes. These adipose compartments are defined as superficial subcutaneous, deep subcutaneous, and internal. Each of these three compartments are further subdivided into abdominal and non-abdominal.
Time Frame: Term plus 6 weeks corrected age
Population: Feed intervention arm
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Unfortified Human Donor Milk | Fortified Human Donor Milk | Preterm Formula
Number analyzed (Participants) | 14 | 5 | 19
Litres | 0.064 (0.023) | 0.061 (0.025) | 0.062 (0.018)

17. Secondary Outcome: Non Adipose Tissue, as Measured by Whole Body MRI at Term Plus 6 Weeks
Description: Non adipose tissue, as measured by whole body MRI, at Term plus 6 weeks. As measured by whole body Magnetic Resonance Imaging (MRI). MR images were acquired using a rapid T1-weighted spin-echo sequence allowing whole body imaging. Images obtained give good contrast between adipose tissue and other tissues, and allows direct measurement of adipose compartment volumes, whole body adipose tissue volume being the sum of these adipose compartment volumes. This volume may be converted to adipose tissue mass on the assumption that the density of adipose tissue is 0.9 g/cm³. Non adipose tissue mass reported here is weight (g) minus whole body adipose mass (g)
Time Frame: Term plus 6 weeks corrected age
Population: Feed intervention arm
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Unfortified Human Donor Milk | Fortified Human Donor Milk | Preterm Formula
Number analyzed (Participants) | 14 | 5 | 19
Grams | 3263.98 (609.89) | 3208.10 (526.21) | 3364.38 (634.07)

18. Secondary Outcome: Blood Quantitative Insulin Sensitivity Check Index (QUICKI)
Description: The quantitative insulin sensitivity check index (QUICKI) is derived using the inverse of the sum of the logarithms of the fasting insulin and fasting glucose:
  1 / (log(fasting insulin μU/mL) + log(fasting glucose mg/dL)). This index correlates well with glucose clamp studies and is useful for measuring insulin sensitivity (IS), which is the inverse of insulin resistance (IR). The higher the value of QUICKI, the higher the measure of insulin sensitivity. Reference ranges for adults, and less so preterm newborns, have not been fully established; values of 0.3 in adults or below are typically associated with insulin resistance or diabetes. In a large cohort of 115 term, normoweight newborns at birth (Gesteiro E. Eur J Pediatr. 2009 Mar;168(3):281-8), mean (95% confidence interval) QUICKI was 0.45 (0.43-0.48)
Time Frame: Measured at 35 weeks Post Menstrual Age
Population: Feed intervention arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Unfortified Human Donor Milk | Fortified Human Donor Milk | Preterm Formula
Number analyzed (Participants) | 13 | 11 | 17
units on a scale | 0.46 (0.09) | 0.42 (0.03) | 0.45 (0.09)

ADVERSE EVENTS:
Time Frame: From period of feed intervention, this is from birth to 35 weeks post menstrual age.
Arm/Group | Unfortified Human Donor Milk | Fortified Human Donor Milk | Preterm Formula
All-Cause Mortality (participants affected / at risk) | 1/35 | 0/34 | 1/34
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/35 | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT01686477/Prot_SAP_000.pdf